CLINICAL TRIAL: NCT05543239
Title: Efficacy and Safety of Transcutaneous Auricular Vagus Nerve Stimulation on Radiotherapy-Related Neuropathic Pain in Patients With Head and Neck Cancers: A Multi-center, Randomized, Double-Blind, Sham-Controlled Trial
Brief Title: Efficacy and Safety of Transcutaneous Auricular Vagus Nerve Stimulation on Radiotherapy-Related Neuropathic Pain
Acronym: RELAX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20220901
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-09

CONDITIONS: Neuropathic Pain; Radiotherapy Side Effect
Keywords: Radiotherapy-Related Neuropathic Pain; Transcutaneous Auricular Vagus Nerve Stimulation; Head and Neck Cancers; Randomized controlled trials
MeSH Terms: conditions — Neuralgia; Radiation Injuries; Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An independent physiotherapist performs vagus nerve stimulation or sham stimulation according to the group envelope; Investigators (physicians) are only responsible for administering medications other than vagus nerve stimulation;Before treatment, all subjects were told that the intensity of this treatment method may not be felt; The therapeutic device is placed in an opaque airtight pouch that is invisible to both the clinician and the patient during use. The control strategy used "transient sham stimulation", which allows for subjects blinding while delivering a true placebo treatment. Data analysts will be blinded to the allocated treatment group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TaVNS (Active Comparator): Patients will receive TaVNS stimulation for 30 minutes, twice a day (between 9:00 to 10:00 and 15:00 to 16:00), for 7 consecutive days. Stimulation pulses (30 Hz frequency, 300 μs pulse width) were generated by a commercial transcutaneous auricular vagus nerve stimulation unit (tVNS 501，Jiangsu, China), and the amplitude was increased to the maximum amount tolerated by the subject without pain, then stimulate for 30 min. All subjects were told that they may or may not feel any sensation from the stimulation, and the unit is packed in an opaque bag throughout the treatment.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation(TaVNS)
- Sham TaVNS (Sham Comparator): Patients will receive sham TaVNS stimulation for 30 minutes, twice a day (between 9:00 to 10:00 and 15:00 to 16:00), for 7 consecutive days. Stimulation unit was active for the first 30s, stimulation pulses (30 Hz frequency, 300 μs pulse width) were generated by a commercial transcutaneous auricular vagus nerve stimulation unit (tVNS 501，Jiangsu, China).Then dropped to zero stimulation during 15s and shut down. All subjects were told that they may or may not feel any sensation from the stimulation, and the unit is packed in an opaque bag throughout the treatment.
  Interventions: Device: Sham Transcutaneous Auricular Vagus Nerve Stimulation(SS)

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation(TaVNS) — Transcutaneous Auricular Vagus Nerve Stimulation (TaVNS) works by stimulating the auricular branches of the vagus nerve (mainly distributed in the concha cavity and conchae) through electrical impulses.Electrodes were placed on the concha of the left ear after cleaning the skin of the concha with a small disposable alcohol pad. Stimulation pulses (frequency 30 Hz, pulse width 300 us) were generated by TaVNS device, the amplitude was increased within 30 seconds to the subject produced a tingling sensation, and then descend within 15 seconds to the maximum tolerable amount without pain. Inform the subject that "target stimulus has been reached", then stimulate for 30 minutes.
  Arms: TaVNS
Device: Sham Transcutaneous Auricular Vagus Nerve Stimulation(SS) — Place electrodes on the concha of the left ear after cleaning the skin of the concha with a small disposable alcohol pad. The same stimulation pulses (30 Hz frequency, 300 us pulse width) were generated by the same device, the amplitude was increased within 30 seconds to the subject produced a tingling sensation, and then ramps down to zero stimulus over 15 seconds. The subjects were told that "the target stimulus has been reached". Patients receive sham stimulation for 30minutes.
  Arms: Sham TaVNS

SUMMARY:
This multi-center, randomized, double-blind, sham-controlled trial aims to investigate the effect and safety of TaVNS in treating radiotherapy-related neuropathic pain.

DETAILED DESCRIPTION:
Radiotherapy-related neuropathic pain(RRNP) is one of the most distressing complications after radiotherapy for head and neck cancers. The prevalence of neuropathic pain in cancer pain patients is as high as 31-45%.Our previous RCT of pregabalin for RRNP showed that nearly 41.6% of patients still did not achieve 30% pain relief even with standard doses of pregabalin. At the same time, drug side effects such as dizziness and obesity are common, and a dose titration process for at least one week is required.Therefore, new treatments that effectively relieve pain and improve quality of life must be explored.

Transcutaneous Auricular Vagus Nerve Stimulation (TaVNS) works by stimulating the auricular branches of the vagus nerve through electrical impulses. Previous studies have shown it can relieve various pains including migraine, cluster headache, musculoskeletal pain with few adverse events. This study plans to evaluate the efficacy of TaVNS versus sham stimulation for relieving RRNP, and assessed its safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥18 years with an estimated survival of at least 5 months;
2. Prior radiotherapy for histologically confirmed cancer ≥ 6 months prior to study entry;
3. Pain for at least 4 weeks with an average intensity of ≥ 4 on an 11-point numeric rating scale (NRS) in the run-in period, and pain locations in accordance with radiated innervated areas, e.g. head, face, neck and arms;
4. Neuropathic pain defined according to clinical history, symptoms, physical signs, and a score ≥ 12 in the Chinese version of Leeds Assessment of Neuropathic Symptoms and Signs questionnaire (LANSS) by two trained and experienced neurology specialists.

Exclusion Criteria:

1. Current diagnosis of tumor recurrence or metastasis and evidence of tumor-associated pain;
2. Patients with non-radiotherapy induced neuropathic pain, e.g. postherpetic neuralgia, diabetes mellitus, HIV infection, spinal cord injury and other neurological disease;
3. Use of carbamazepine, gabapentin, pregabalin, TaVNS or transcranial magnetic stimulation within the last 30 days prior to study entry;
4. Other ongoing treatment for neuropathic pain, including antidepressants with norepinephrine and serotonin reuptake inhibition, calcium channel α2-δ ligands and other anticonvulsant medications, and topical lidocaine;
5. Concomitant medication that may cause an adverse interaction with pregabalin, including sedative (e.g., benzodiazepines);
6. Significant renal impairment: plasma creatinine>1.5mg/ml, creatinine clearance < 60 mL/min;
7. History of anaphylactic response to pregabalin;
8. Ulceration of the auricle skin; Diagnosis of mental illness, peptic ulcer,AV III degree block, heart rate< 50/min, heart rate corrected QT interval > 450ms;
9. Patients with cardiac pacemakers or implanted ECG monitoring equipment;
10. Evidence of severe systemic diseases;
11. Subjects with any other condition which, in the investigator's judgment might interfere the outcome of the study;
12. Refuse to provide written informed consent;
13. Cognitive function and language skills are insufficient to complete study questionnaires;
14. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to day 7 with respect to pain intensity based on the NRS. | Day 7
  The primary outcome of this trial is to evaluate the change from baseline to Day 7 with respect to pain intensity based on the NRS, which evaluates the average pain in the last 24 hours from "0" indicating "No Pain" to "10" indicating "Pain as bad as you can imagine".

SECONDARY OUTCOMES:
Change from baseline to week 16 with respect to pain intensity based on the NRS. | week 16
  The primary outcome of this trial is to evaluate the change from baseline to Day 7 with respect to pain intensity based on the NRS, which evaluates the average pain in the last 24 hours from "0" indicating "No Pain" to "10" indicating "Pain as bad as you can imagine".
BPI-SF | day 7, week 16
  The Chinese version of Brief Pain Inventory (Short-Form) is used to assesses pain severity and inference, which has been widely used in neuropathic pain. The Pain severity score is assessed as mean of the four pain items (i.e., pain at its worst, least, average, and now)29. Functional inference is measured by the BPI Interference in 7 items, which includes General activity, Mood, Walking ability, Work, Social relations, Sleep and Life enjoyment. Each item is scored on a 10-point scale. Lower scores indicate alleviative functional interference.
POMS-SF | day 7, week 16
  The Chinese version of short form of the Profile of Mood States (POMS-SF) has been recommended as core outcome measures of emotional functioning in chronic pain clinical trials. It's a 30-item scale to evaluate patients' mood states, including 5 negative mood states (Tension-anxiety, Depression-Dejection, Anger-Hostility, Fatigue-Inertia, Confusion-Bewilderment) and 1 positive mood state (Vigor-Activity).Lower scores indicate alleviative mood disturbance in all fields except the positive one.
WHOQOL-BREF | day 7, week 16
  The Chinese version of WHOQOL-BREF is a brief version of The World Health Organization Quality of Life (WHOQOL), which has been widely used in clinical studies on cancer and neuropathic pain. In the questionnaire, a total of 26 items assess 4 domains of quality of life, including physiology, psychology, social relationship and environment. Lower scores correspond to poorer quality of life.
FACIT-F | day 7, week 16
  The Chinese version of the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) is widely used to assess various chronic disease-related fatigue states. The FACIT-F is a self-report scale. It comprises 13 items with five-point response options from 0 to 4. Except for items An5 and An7, which are forward scoring, all other items are reverse scoring. The total score ranges from 0 to 52, with a higher total score representing less fatigue.
PGIC | day 7, week 16
  The Patient Global Impression of Change (PGIC) is self-evaluation of the patient's overall change on a 7-point scale (1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; 7 = very much worse), and is obtained at the end of the study. Treatment success is defined as "much" or "very much" improved. The PGIC question will ask: "With respect to your overall radiotherapy-related neuropathic pain symptoms, how will you describe yourself now compared to immediately before starting study medication?"
CGIC | day 7, week 16
  The Clinical Global Impression of Change (CGIC) is single item questionnaire that asks the investigator to evaluate the subject's overall symptom change on a 7-point scale (1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; 7 = very much worse), and is obtained at the end of the study. Treatment success is defined as "much" or "very much" improved. The CGIC question will ask: "With respect to the subject's overall radiotherapy-related neuropathic pain symptoms, how will you describe him (or her) now compared to immediately before starting study medication?"
Serum Inflammatory Factors | day 7
  The serum inflammatory factors including: serum tumor necrosis factor-α (TNF-α) level; serum interleukin-1beta (IL-1β) level; serum interleukin-6 (IL-6) level; serum interleukin-10 (IL-10) level.Whole blood was centrifuged, serum was then stored at -80°C. The inflammatory factors were detected by ELISA in the laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Yamei Tang, M.D.;PHD., Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (4):
- China (4):
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Department of Nasopharyngeal Carcinoma, Sun Yat-Sen University Cancer Center, Guangzhou
  - Department of Nasopharyngeal Carcinoma, The Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou
  - Department of Neurology, The Affiliated Brain Hospital of Guangzhou Medical University, Guangzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zuo X, Xu Y, Li S, Jiang J, Wang J, Zhu Y, Pan D, Li H, Chen Y, Chen Y, Rong X, Zheng D, Lu K, Mai H, Chen M, Chen P, Li J, Simone CB, Chua MLK, Li Y, Shen Q, Xiao S, Tang Y. Efficacy and safety of transcutaneous auricular vagus nerve stimulation plus pregabalin for radiotherapy-related neuropathic pain in patients with head and neck cancer (RELAX): a phase 2 randomised trial. EClinicalMedicine. 2025 Jul 12;86:103345. doi: 10.1016/j.eclinm.2025.103345. eCollection 2025 Aug. PMID 40697962
- [Derived] Zuo X, Li Y, Rong X, Yang X, Zhu Y, Pan D, Li H, Shen QY, Tang Y. Efficacy of transcutaneous auricular vagus nerve stimulation on radiotherapy-related neuropathic pain in patients with head and neck cancers (RELAX): protocol for a multicentre, randomised, double-blind, sham-controlled trial. BMJ Open. 2023 Sep 20;13(9):e072724. doi: 10.1136/bmjopen-2023-072724. PMID 37730386